CLINICAL TRIAL: NCT03700528
Title: The Development of Contextual Cognitive Behavioural Approach to Painful Diabetic Neuropathy: A Feasibility Trial
Brief Title: The Development of Contextual Cognitive Behavioural Approach to PDN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Diabetes UK (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS ID 224386
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus; Painful Diabetic Neuropathy
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Neuropathies | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: The psychological treatment which we will use is called Acceptance and Commitment Therapy (ACT). The ACT treatment includes treatment processes of acceptance, cognitive defusion, mindfulness, and values-based action. Methods will include practice to deal with painful experiences, to improve awareness, to identify and work on goals, and to better stick to commitments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): This is a single-cohort ACT based intervention.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — The process will involve, two, brief, one-to-one contact sessions, one at the beginning and one at the end of the intervention, in a way that is convenient for participants, including Skype, phone, or face to face in person. Following the first one-to-one session there will be eight short online sessions, about 20-30 minutes each. Participants will also be asked to complete some tasks between the sessions, in particular to record their progress briefly and any changes at their medication (i.e. type of drug, dose) in a diary weekly so that they can keep track of your developing skills.

SUMMARY:
Diabetes mellitus (DM) is highly prevalent, and a significant public health problem. Approximately 25-30% of all individuals with DM develop painful diabetic neuropathy (PDN). PDN is considered a complex, multi-dimensional condition, possibly affecting the physical and mental health of the individual. PDN is usually described as a sense of burning, stabbing, aching and/or pricking mainly affecting areas like toes, legs, and feet and physically interfering with mobility, sleep, mood, and overall quality of life. This condition represents both a significant problem in its own right and a useful condition in which to test treatments that may offer wider benefits for neuropathic pain conditions in general.

A relatively new and promising approach to chronic pain, within the wider range of cognitive and behavioural approaches, is Acceptance and Commitment Therapy (ACT). ACT is a form of Cognitive Behavioural Therapy (CBT) that focuses specifically on increasing psychological flexibility. Psychological flexibility is the capacity to change or continue with a behaviour, depending on which is more effective, according to one's goals and what the current situation affords. Psychological flexibility in turn includes processes of acceptance, values-based action, and other processes related to mindfulness. There are no published studies of ACT for individuals with PDN, and the limited available evidence indicates that a CBT-based intervention like ACT has the potential to reduce pain in people with PDN. People with PDN have clear treatment needs. While ACT may help them, little is known directly about the relevance of different components of ACT for this condition or about how to customise it for them. The proposed research aims to conduct a small feasibility trial which will pilot test a psychological treatment for PDN and assess the feasibility, acceptability and effectiveness of such a treatment.

DETAILED DESCRIPTION:
People with diabetes often experience a type of pain called Painful Diabetic Neuropathy (PDN). PDN is described as a stabbing, burning, pricking, or aching sensation affecting the toes, feet, and legs. This type of pain can interfere with walking, sleep, mood and overall quality of life. Although medication may offer some short-term improvement in this pain, this is a chronic condition for the majority of the patients and the pain typically remains a problem. Our research team aims to assess the acceptability and potential benefits of a psychological treatment for people with PDN.

The intervention is a tailored ACT-based self-management intervention which will be delivered online. The purpose of this intervention is to improve participant daily functioning via increased psychological flexibility. The development of the PDN ACT-based intervention involved a multidisciplinary team of psychologists, health professionals and diabetes specialists.

The ACT treatment package will embrace the core treatment processes of acceptance, cognitive defusion, mindfulness, and values-based action. Methods will include practice in contacting painful experiences, experiential cognitive methods to promote awareness, exercises similar to mindfulness, methods to increase one's the role of goals and values in patient choice, and to help people flexibly stick to commitments.

The process will involve, two brief direct one-to-one contact sessions, one at the beginning and one at the end of the intervention, with convenient means according to each participant, as for example Skype, phone or face to face. Following the first one-to-one session there will be 8 short online sessions, with a duration of 20-30 minutes each. In accordance with ACT principles, participants will be encouraged to complete tasks between the online sessions. Particularly, they will be asked to write on a diary weekly, which will include ratings for openness, awareness and engagement. Within the diary we will also ask participants to note changes, in medication, if any, and if the data is sufficient and relevant we will include them in the final analysis. The completion of these tasks has been found to be predictive of CBT outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years.
* Confirmed diagnosis of diabetes.
* Presence of painful diabetic neuropathy.
* Have full verbal and written proficiency in English.
* Willingness and ability to take part.
* Have computer literacy.

Exclusion Criteria:

* Not understanding verbal explanation or written information in English.
* Suffering from neuropathy due to other causes than diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Committed Action Questionnaire (CAQ-8) | 8 weeks
  The CAQ-8 is an eight-item measure of committed action, a facet of PF. Committed action is the ability to persist with actions that are guided by goals, including when this runs into discouraging experiences and to change these actions when they are shown to be ineffective. Responses to the items were rated from 0 (never true) to 6 (always true). Out of the eight items four are positively keyed and four negatively keyed.

SECONDARY OUTCOMES:
Cognitive Fusion Questionnaire (CFQ-7) | 8 weeks
  The CFQ-7 offers a psychometrically sound measure of cognitive fusion. 16 Cognitive fusion refers to a domination of cognitive influence over direct experiential influence on behavior, and a lack of separation between the content of the thoughts and the situations or people to which they refer. Cognitive defusion, on the other hand, is the ability to see thoughts as just thoughts, and not as essential reflections of events as they are directly experienced. CFQ-7 consists of 7-items rated on a 0 (never true) to 7 (always true) point scale. An early version of the CFQ has been validated in chronic pain sample.
Chronic Pain Acceptance Questionnaire (CPAQ-8) | 8 weeks
  The CPAQ-8 is a validated questionnaire which measures acceptance of chronic pain. It includes engagement in activities while experiencing pain and willingness to experience pain without trying to control or avoid it. CPAQ-8 is based on the 20-item questionnaire and has been validated 12. Items are rated on a scale from 0 (never true) to 6 (always true). Higher scores reflect greater acceptance of pain.
Douleur neuropathique 4 (DN4) | 8 weeks
  Presence of neuropathic pain was assessed with a screening measure called DN4. It consists of interview questions and physical tests and has also been validated as a self-reported measure. It has a specificity of 83% and sensitivity of 90%.
Pain Scale | 8 weeks
  Pain intensity and distress were assessed through four questions using 0 (no pain) to 10 (worst possible pain) numerical ratings of pain. Participants were asked to rate their pain right now and in the past week, and how distressing is their pain right now and in the past week.
Patient Health Questionnaire (PHQ-9) | 8 weeks
  The PHQ-9 is a reliable and validated measure used as an index for depression severity. It includes 10-items based on DSM-IV. The nine items that reflect severity of depression symptoms area each rated on a scale from 0 (not at all) to 4 (nearly every day). The last item is a measure of impact of depression and is rated from 'not difficult at all' to 'extremely difficult'. The higher score indicates higher levels of depression severity.
Self Experiences Questionnaire (SEQ) | 8 weeks
  The SEQ is a 15-item self-report measure of self-as-context (SAC), within the PF model. This "contextual self" is defined as a sense of self that is not based upon self-evaluations and is separate from one's thoughts and feelings. This could also be referred as, taking a point of view on one's psychological experiences, or as "perspective taking". All items are rated on a scale from 0 (never true) to 6 (always true). All items are positively keyed, and higher scores indicate higher PF.
Work and Social Adjustment Scale (WSAS) | 8 weeks
  The WSAS is a five-item, reliable and validated, self-report measure of impairment in work and social functioning, or as we label in here, "functional impairment". Each item is rated from 0 (no impairment) to 8 (very severe impairment). WSAS items refer to work, home management, social and private leisure, and relationships.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - St Thomas' NHS Foundation Trust (Diabetes Clinic), London
  - Guy's hospital NHS Foundation Trust (Diabetes Clinic), London

IPD SHARING:
Plan to Share IPD: No
King's College London (KCL) and Guy's and St Thomas' NHS Foundation trust (GSTT) are the co-sponsors for this study based in the United Kingdom. They will be using information from participants in order to undertake this study and will act as the data controller for this study. This means that they are responsible for looking after participants' information and using it properly. King's College London and Guy's and St Thomas' NHS Foundation trust will keep identifiable information about participants for 7 years after the study has finished. Participants rights to access, change or move information are limited, as KCL and GSTT need to manage participants information in specific ways in order for the research to be reliable and accurate. If participants withdraw from the study, KCL and GSTT will keep the information about them that have already been obtained. To safeguard participants rights, KCL and GSTT will use the minimum personally-identifiable information possible.